CLINICAL TRIAL: NCT04968197
Title: Vestibular Intervention Via Portable Electrical Stimulator (VIPES)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gaurav N. Pradhan, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-005284
Record Dates: First submitted 2021-07-07; First posted 2021-07-20 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Balance Disorder
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Stochastic Vestibular Stimulation (SVS) Condition (Experimental): Subjects will perform standard clinical testing for balance and gait while wearing the Vestibular Intervention via Portable Electrical Stimulator (VIPES) system. The SVS device will be active throughout the testing at the respective current levels (i.e., 0.2mA to 1 mA at 0.2 mA increments).
  Interventions: Device: Vestibular Intervention via Portable Electrical Stimulator (VIPES) system
- Control Condition (No Intervention): Subjects will perform standard clinical testing for balance and gait without SVS

INTERVENTIONS:
Device: Vestibular Intervention via Portable Electrical Stimulator (VIPES) system — A small, lightweight device able to deliver stochastic vestibular stimulation (SVS) using a comfortable electrode set on the back of the head as well as other proven modes of galvanic vestibular stimulation (GVS) related vestibular correction when required to mitigate motion sickness or provide auxiliary vestibular cueing.
  Arms: Stochastic Vestibular Stimulation (SVS) Condition

SUMMARY:
The purpose of this study is to develop a vestibular interventional approach using stochastic vestibular stimulation (SVS) through a small, lightweight device, and a comfortable electrode set on the back of the head that stimulates the vestibular system and produces immediate improvements in balance, gait, and overall vestibular function for patients will balance disorder.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to consent to participate themselves.
* Must be able to attend in-person sessions at the Mayo Aerospace Medicine and - Vestibular Research Laboratory in Scottsdale, AZ.
* No racial/ethnic groups will be excluded.
* All participants must be fluent speakers of English.

Exclusion Criteria:

* Presence of peripheral vestibulopathy (cleared by Dix-Hallpike, vHIT as part of clinical evaluation).
* Women who are pregnant.
* Inability to complete testing (e.g., severe symptom burden, inability to stand unassisted).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav N Pradhan, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 23 participants were enrolled to receive all interventions; however, the order the intervention was received was randomized. All subjects completed all study visits/interventions.
Groups:
- All Participants Stochastic Vestibular Stimulation (SVS) and Control Condition: All subjects will perform standard clinical testing for balance and gait without SVS and while wearing the Vestibular Intervention via Portable Electrical Stimulator (VIPES) system. The SVS device will be active throughout the testing at the respective current levels (i.e., 0.2mA to 1 mA at 0.2 mA increments).
  Vestibular Intervention via Portable Electrical Stimulator (VIPES) system: A small, lightweight device able to deliver stochastic vestibular stimulation (SVS) using a comfortable electrode set on the back of the head as well as other proven modes of galvanic vestibular stimulation (GVS) related vestibular correction when required to mitigate motion sickness or provide auxiliary vestibular cueing.
Period: Overall Study
Arm/Group | All Participants Stochastic Vestibular Stimulation (SVS) and Control Condition
Started | 23
Control Condition | 23
0.33mA Stochastic Vestibular Stimulation | 23
0.67mA Stochastic Vestibular Stimulation | 23
1mA Stochastic Vestibular Stimulation | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants Stochastic Vestibular Stimulation (SVS) and Control Condition
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Balance Performance
Description: Change in balance performance during balance testing by measuring the center of gravity sway (degrees per second) across tested levels of GVR amplitude and control condition.
Time Frame: Through study completion, approximately 1.5 hours
Measure: Mean (Standard Deviation); unit: degrees per second
Groups:
- Control Condition: Subjects will perform standard clinical testing for balance and gait without stochastic vestibular stimulation (SVS)
- 0.33 Milliamps (mA) Stochastic Vestibular Stimulation (SVS) Condition; 0.67 Milliamps (mA) Stochastic Vestibular Stimulation (SVS) Condition; 1 Milliamps (mA)Stochastic Vestibular Stimulation (SVS) Condition: Subjects will perform standard clinical testing for balance and gait while wearing the Vestibular Intervention via Portable Electrical Stimulator (VIPES) system. The SVS device will be active throughout the testing at the respective current levels (i.e., 0.2mA to 1 mA at 0.2 mA increments).
  Vestibular Intervention via Portable Electrical Stimulator (VIPES) system: A small, lightweight device able to deliver stochastic vestibular stimulation (SVS) using a comfortable electrode set on the back of the head as well as other proven modes of galvanic vestibular stimulation (GVS) related vestibular correction when required to mitigate motion sickness or provide auxiliary vestibular cueing.
Arm/Group | Control Condition | 0.33 Milliamps (mA) Stochastic Vestibular Stimulation (SVS) Condition | 0.67 Milliamps (mA) Stochastic Vestibular Stimulation (SVS) Condition | 1 Milliamps (mA)Stochastic Vestibular Stimulation (SVS) Condition
Number analyzed (Participants) | 23 | 23 | 23 | 23
degrees per second
  Eye Open Firm Surface | 0.52 (0.84) | 0.42 (0.34) | 0.51 (0.79) | 0.48 (0.57)
  Eye Closed Firm Surface | 0.63 (0.81) | 0.55 (0.69) | 0.73 (1.19) | 0.58 (0.69)
  Eye Open Foam Surface | 0.91 (1.12) | 0.73 (0.58) | 0.87 (0.77) | 0.76 (0.47)
  Eye Closed Foam Surface | 1.36 (0.97) | 1.49 (1.58) | 1.47 (1.23) | 1.47 (1.32)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately an hour and a half on all participants.
Arm/Group | Control Condition | 0.33 Milliamps (mA) Stochastic Vestibular Stimulation (SVS) Condition | 0.67 Milliamps (mA) Stochastic Vestibular Stimulation (SVS) Condition | 1 Milliamps (mA)Stochastic Vestibular Stimulation (SVS) Condition
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT04968197/Prot_SAP_000.pdf